CLINICAL TRIAL: NCT05172947
Title: Impact of Resveratrol and Pharmaceutical Care on Diabetes Mellitus and Its Neuropathic Complication
Brief Title: Effect of Resveratrol and Pharmacist Intervention on Diabetes Mellitus and Its Neuropathic Complication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sulaimani (Other)
Responsible Party: Principal Investigator, Bushra Hassan Marouf, Assistant Professor at Pharmacology and Toxicology Department, University of Sulaimani
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: University of Sulaimani
Record Dates: First submitted 2021-11-30; First posted 2021-12-29 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Diabetic Neuropathies
Keywords: Diabetic neuropathy; Neuropathic pain; pharmaceutical care; Resveratrol
MeSH Terms: conditions — Diabetic Neuropathies; Neuralgia | interventions — Resveratrol; Pharmaceutical Services

STUDY DESIGN:
Intervention Model Description: Eligible patients assigned to either conventional hypoglycemic drugs without pharmaceutical care, or conventional hypoglycemic drugs accompanied with pharmacist interventions or patients will receive resveratrol 500 mg capsules orally once daily with their regular hypoglycemic drugs or resveratrol 500 mg capsule orally along with their regular hypoglycemic drugs for a period of three months, accompanied with pharmacist interventions.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A prospective triple blind randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Resveratrol (Active Comparator): Interventional group, participants in this group are receiving Resveratrol 500mg capsule once daily for 3 months.
  Interventions: Drug: Resveratrol
- Placebo (Placebo Comparator): Non-interventional group, participants are receiving only Placebo once daily for 3 months.
  Placebo formulated as capsule match the color and size of the active comparator,
  Interventions: Drug: Placebo
- Resveratrol plus Pharmaceutical care (Other): Interventional group, participants in this group are receiving Resveratrol 500mg capsule once daily for 3 months with pharmaceutical care.
  Interventions: Other: Resveratrol plus Pharmaceutical care
- Placebo with pharmaceutical care (Other): Interventional group, participants are receiving placebo along with pharmaceutical care for 3 months.
  Interventions: Other: Placebo+Pharmaceutical care

INTERVENTIONS:
Drug: Resveratrol — This group received resveratrol with the conventional therapy
  Arms: Resveratrol
Drug: Placebo — This group received placebo with the conventional therapy
  Arms: Placebo
Other: Resveratrol plus Pharmaceutical care — This group received Resveratrol with Pharmaceutical care in addition to the conventional therapy
  Arms: Resveratrol plus Pharmaceutical care
Other: Placebo+Pharmaceutical care — This group received placebo with Pharmaceutical care in addition to the conventional therapy
  Arms: Placebo with pharmaceutical care

SUMMARY:
Management of symptoms associated with diabetic neuropathy is a difficult issue for clinicians since it usually does not respond to standard analgesics. Resveratrol is a naturally occurring plant-derived, polyphenolic compound, it exerts pleiotropic activity. The investigators believed that the implementation of multidisciplinary approaches including pharmacotherapy and provision of healthcare professional services such as pharmacist intervention are needed for alleviation of diabetic associated neuropathy.Therefore, the hypothesis of the present protocol is that the administration of resveratrol and/or provision of pharmaceutical care in patients with diabetic neuropathy might be of value in improving quality of life and managing diabetic neuropathic pain.The study is designed as a four-arm randomized, placebo-controlled clinical trial. Group one will be given only conventional hypoglycemic drugs. Group two patients will receive conventional hypoglycemic drugs accompanied by pharmacist interventions. Group three; patients will receive resveratrol 500 mg orally once daily after meals for three months, in addition to their regular hypoglycemic drugs. Group four; patients will receive resveratrol 500 mg orally once daily after meals along with their regular hypoglycemic drugs for a period of three months, accompanied by pharmacist interventions. Neuropathic pain will be measured by various neuropathic pain assessment tools. Nerve conduction studies will be performed to assess the effect of interventional therapy. The expected outcome will be the improvement of diabetic neuropathy associated symptoms along with glycemic status.

DETAILED DESCRIPTION:
* Diabetic neuropathy is the most common microvascular complication of diabetes, resulting from prolonged periods of hyperglycemia, damaging fragile nerve fibers and the walls of their blood vessels.
* Despite clinical developments in the treatment of diabetes complications, especially diabetic neuropathy, it still remains a clinical challenge with no effective solution.
* Conventional therapies such as anti-epileptics, opioid analgesics, and antidepressants for the treatment of neuropathic pain are quite challenging due to their serious adverse effects.
* There is a need to investigate novel effective and safe options.
* Recently, polyphenols have also been introduced as potential neuroprotective agents in diabetes.
* Alleviation of the symptoms associated with diabetic neuropathy and exerting preventive measures to halt the emergence of neuropathy complications are crucial priorities, and this requires multidisciplinary approaches including pharmacotherapy and provision of healthcare professional services such as pharmacist intervention.
* Aim of the study: to evaluate the effects of resveratrol and pharmaceutical care on the severity of diabetic neuropathy and improvement in the quality of life of diabetic patients.
* Study design: four-arm randomized, double-blind, placebo-controlled clinical trial.
* Interventions:Therapeutic intervention and Pharmacist intervention.
* Number of participants = 120
* Number of groups = 4 groups each of 30 patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with pain due to bilateral peripheral neuropathy caused by type 2 diabetes mellitus.
* HbA1c of greater than 7%
* The daily pain must be present for at least 6 months, and the diagnosis will be confirmed by a score >4 on the Michigan Neuropathy Screening Instrument (MNSI), Douleur Neuropathique 4 (DN4). The severity of pain when evaluated for the past 24 was ≥4 on the 10 cm Visual Analogue Scale (VAS) at baseline without the use of analgesic for 48 hours.

Exclusion Criteria:

* Older subjects with high risks of cardiovascular diseases,
* Pregnant or breastfeeding,
* Having a prior renal transplant or current renal dialysis,
* Patients have a diagnosis of major depressive disorder, generalized anxiety disorder, heavy alcohol drinkers,
* Significant hepatic or renal disease,
* Patients on antioxidant therapy, or pentoxyphylline within the last month.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-12-05 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
visual analog scale (VAS) | up to 3 months
  to assess neuropathic pain, VAS scale ranges between 0-10 , 0 indicates no pain while 10 indicates severe pain.
Douleur Neuropathique 4 questionnaire (DN4) | up to 3 months
  to assess the severity of diabetic peripheral neuropathy.
The Michigan Neuropathy Screening Instrument (MNSI) | up to 3 months
  to assess the severity of diabetic peripheral neuropathy
Electroneurography | up to 3 months
  Motor nerve conduction velocity (m/s), sensory nerve conduction velocity(m/s) will be measured using surface electrodes.
Assessment of Quality of Life | up to 3 months
  using the RAND-36 health survey questionnaire
Serum neopterin levels | up to 3 months
  biochemical marker for peripheral neuropathy

SECONDARY OUTCOMES:
The mean change in fasting blood glucose | up to 3 months
  to assess glycemic status
Mean change of glycated hemoglobin (HbA1c)-mmol/l | up to 3 months
  to assess glycemic status
Measurement of serum level of LDL, cholesterol, HDL, Triglyceride | up to 3 months
  to assess the effect of the interventions on metabolic changes

CONTACTS AND LOCATIONS:
Overall Officials: Bushra Marouf, PhD, Principal Investigator — Department of Pharmacology and Toxicology-College of Pharmacy-University of Sulaimani
Locations (1):
- College of Pharmacy-University of Sulaimani, Sulaymānīyah, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azmi S, ElHadd KT, Nelson A, Chapman A, Bowling FL, Perumbalath A, Lim J, Marshall A, Malik RA, Alam U. Pregabalin in the Management of Painful Diabetic Neuropathy: A Narrative Review. Diabetes Ther. 2019 Feb;10(1):35-56. doi: 10.1007/s13300-018-0550-x. Epub 2018 Dec 18. PMID 30565054
- [Background] Collins C, Limone BL, Scholle JM, Coleman CI. Effect of pharmacist intervention on glycemic control in diabetes. Diabetes Res Clin Pract. 2011 May;92(2):145-52. doi: 10.1016/j.diabres.2010.09.023. Epub 2010 Oct 20. PMID 20961643
- [Background] Elbarbary NS, Ismail EAR, El-Hilaly RA, Ahmed FS. Role of neopterin as a biochemical marker for peripheral neuropathy in pediatric patients with type 1 diabetes: Relation to nerve conduction studies. Int Immunopharmacol. 2018 Jun;59:68-75. doi: 10.1016/j.intimp.2018.03.026. Epub 2018 Apr 6. PMID 29627577
- [Background] Naseri R, Farzaei F, Fakhri S, El-Senduny FF, Altouhamy M, Bahramsoltani R, Ebrahimi F, Rahimi R, Farzaei MH. Polyphenols for diabetes associated neuropathy: Pharmacological targets and clinical perspective. Daru. 2019 Dec;27(2):781-798. doi: 10.1007/s40199-019-00289-w. Epub 2019 Jul 27. PMID 31352568
- [Background] Eid S, Sas KM, Abcouwer SF, Feldman EL, Gardner TW, Pennathur S, Fort PE. New insights into the mechanisms of diabetic complications: role of lipids and lipid metabolism. Diabetologia. 2019 Sep;62(9):1539-1549. doi: 10.1007/s00125-019-4959-1. Epub 2019 Jul 25. PMID 31346658